CLINICAL TRIAL: NCT06344754
Title: The Effect of Family Planning Education Delivered With the Gamification Method on the Knowledge and Attitudes of University Students
Brief Title: Gamification in Family Planning Education: Impact on University Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, Özlem Ülkü BULUT, PhD Lecturer, Lokman Hekim University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: gamifiedfamilyplanning
Record Dates: First submitted 2024-03-22; First posted 2024-04-03 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Gamification; Reproductive Health; Family Planning; Students
Keywords: gamification; family planning; university students; reproductive health

STUDY DESIGN:
Intervention Model Description: pre-test and post-test interventional study
Masking Description: the person doing the statistical analysis will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gamified Family Planning Education (Experimental): Family planning training will be provided to university students through gamification.
  Interventions: Behavioral: Gamified education

INTERVENTIONS:
Behavioral: Gamified education — Assessment of students' attitudes toward family planning using the Family Planning Attitude Scale, administered as pre-test and post-test to evaluate changes following the educational intervention.

SUMMARY:
More than 3 billion of the worlds population are young people under the age of 25. According to WHO data, one million girls under the age of 15 give birth each year, mostly in low- and middle-income countries, and 3 million adolescent girls between the ages of 15 and 19 are exposed to unsafe abortions. Failure to meet the family planning needs of young people in a timely, adequate and appropriate manner can have significant public health impacts. According to World Health Statistics, the global birth rate for girls between 15 and 19 years of age is 49 out of 1000, and early pregnancy and childbirth can lead to serious health and social problems. In addition, this age group does not have sufficient information about pregnancy and its complications, and their access to and utilization of health services is low. Inadequacies in the education of adolescents on sexual issues and sociocultural differences further increase the sexual and reproductive health risks of young people in the university period. Information and services that will enable individuals to understand their sexuality and help them protect themselves from sexual risks should be provided specifically for that age. Therefore, it is important for young people to know family planning methods. In this study, it was aimed to examine the effect of family planning education to be given with gamification method, which is different from the classical method in the literature, on the knowledge and attitudes of university students.

DETAILED DESCRIPTION:
Location of the research: The research will be conducted with students studying at Lokman Hekim University.

Time of the research: The research will be conducted in the fall semester of the 2023-2024 academic year.

Population, sample and research group: The population of the study will consist of students studying in the midwifery department. Students who agree to participate in the research will constitute the sample of the research.

Type of research: The research was planned as a one-group pretest-posttest quasi-experimental type with the aim of evaluating the effect of the education given with gamification method on the knowledge and attitudes of university students.

ELIGIBILITY:
Inclusion Criteria:

* not having received family planning training before
* having a smartphone

Exclusion Criteria:

* to have received family planning training before

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Knowledge and attitude towards family planning | The measurement tools were administered one week before the training and one month after the training was completed. The study was completed in 5 weeks.
  The research is a one-group pretest-posttest design study conducted to evaluate the effect of gamified education on university students' knowledge and attitudes toward family planning. The purpose and procedure of the study were explained to all eligible students, and informed consent was obtained prior to participation. An introductory information form and the Family Planning Attitude Scale (FPAS) were administered as a pre-test to the students who agreed to participate.
  The Family Planning Attitude Scale is a 5-point Likert-type scale consisting of 34 items, with total scores ranging from 34 to 170. Higher scores indicate more positive attitudes toward family planning, while lower scores reflect more negative attitudes.
  Following the pre-test assessment, each student included in the study group received an online gamified family planning training session delivered by the researchers using Web 2.0 tools. The training lasted approximately 20 minutes per participant.

CONTACTS AND LOCATIONS:
Locations (1):
- Lokman Hekim University, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The study was planned as a one-group pretest-posttest quasi-experimental study with the aim of evaluating the effect of gamification education on the knowledge and attitudes of university students.